CLINICAL TRIAL: NCT04005469
Title: A Phase I/II Study Evaluating the Preliminary Safety and Efficacy of Treprostinil (Remodulin®) In Reducing Ischemia-Reperfusion Injury During De Novo Adult Kidney Transplantation
Brief Title: Safety and Efficacy of Treprostinil (Remodulin®) In Reducing Ischemia-Reperfusion Injury During Kidney Transplantation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Rhode Island (Other); United Therapeutics (Industry)
Responsible Party: Principal Investigator, Reginald Gohh, MD, Rhode Island Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 974570-5
Record Dates: First submitted 2019-06-14; First posted 2019-07-02 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Ischemia Reperfusion Injury; Delayed Graft Function
Keywords: Ischemia-reperfusion injury; kidney transplantation; prostacyclin; treprostinil; delayed graft function
MeSH Terms: conditions — Reperfusion Injury; Delayed Graft Function | interventions — treprostinil

STUDY DESIGN:
Intervention Model Description: Treprostinil will be administered intravenously by a standard 3 + 3 dose-escalation approach. The first three patients will receive a starting rate of 1.25 ng/kg/min and if all three patients safely tolerate the first dose, the next three patients will receive a dose of 2.5 ng/kg/min. If any patients experience side effects, additional patients will receive the previous lower dose. This dosing model will be followed until a target dose of 15 mg/kg/min is achieved or if it is medically determined that side effects prevent dose escalation.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trepostinil (Experimental): Treprostinil (Remodulin) will be administered IV by a standard 3 + 3 dose-escalation approach. This dosing model will be followed until a target dose of 15 mg/kg/min is achieved or if it is medically determined that side effects prevent dose escalation. IV infusion will commence approximately 2-3 hours before transplantation of the kidney graft and will continue for approximately 48 hours after completion of surgery, unless hemodynamic changes or tolerability require discontinuation of treprostinil.
  Interventions: Drug: Treprostinil

INTERVENTIONS:
Drug: Treprostinil — Treprostinil (Remodulin) will be administered IV by a standard 3 + 3 dose-escalation approach. This dosing model will be followed until a target dose of 15 mg/kg/min is achieved or if it is medically determined that side effects prevent dose escalation. IV infusion will commence approximately 2-3 hours before transplantation of the kidney graft and will continue for approximately 48 hours after completion of surgery, unless hemodynamic changes or tolerability require discontinuation of treprostinil.
  Other Names: Remodulin®

SUMMARY:
The objectives of this study are to test the preliminary safety and efficacy of a two-day peri-operative course of treprostinil in reducing ischemia-reperfusion injury in adult patients receiving a deceased donor kidney transplantation. Treprostinil, a prostacyclin analog, is expected to facilitate the restoration of blood supply to the revascularized kidney graft via its vasodilatory actions, well characterized protective effects, and longer elimination half-life. These properties and actions of treprostinil make it a strong drug candidate to reduce kidney graft dysfunction during kidney transplantation. An anticipated 20 participants undergoing deceased donor kidney transplant will be hospitalized and intensively monitored during an entire two-day Treatment Phase. An IV infusion using a dedicated central venous line will be used to administer treprostinil commencing approximately 2-3 hours before transplantation of the kidney graft and will continue for approximately 48 hours after completion of the transplant surgery. The primary endpoints include the safety and efficacy of treprostinil, with secondary endpoints including the evaluation of both biochemical and clinical endpoints post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients who will receive a deceased donor kidney aged 18 to 65 (inclusive) and are currently on the active transplant list at RIH.
2. Documentation of a diabetes diagnosis as evidenced by one or more clinical features consistent will be noted for all patients.
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Under the age of 18 years
2. Difficult venous access
3. BMI > 40 kg/m2
4. Patients with severe clinical gastroparesis as determined by repeated vomiting
5. Prior GI surgery except for cholecystectomy, appendectomy, or Nissen fundoplication
6. Known or history of inflammatory bowel disease or bezoars
7. History of diverticulitis, diverticular stricture, and other intestinal strictures
8. Be receiving any investigational drug other than treprostinil or participating in any other investigational study
9. Be receiving any prostanoid therapy to treat portopulmonary hypertension
10. Have any known hypersensitivity to prostaglandins, prostacyclin or treprostinil
11. Have had a failed kidney transplant within the previous 180 days
12. Be receiving any non-standard immunosuppression protocol or other non-standard treatment that could affect interpretation of the study results
13. Those with significant cardiovascular disease including treatment with inotropes
14. If female, be pregnant or nursing (confirmed by urine test)
15. Presence of a condition or abnormality that in the opinion of the Investigators that would compromise the safety of the patient or the quality of the data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine (SCr) | Day 1-7
  Primary efficacy assessment will include the cGFR using SCr during the first seven days post transplantation.

SECONDARY OUTCOMES:
INR | Day 7
  biochemical end point
Urine output | Day 7
  biochemical end point
Primary graft non-function; kidney failure | Day 30
  dialysis, death or re-transplantation
Delayed graft function | Day 30
  use of dialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided